CLINICAL TRIAL: NCT07152925
Title: The Impact of Beta-band Transcranial Alternating Current Stimulation (tACS) on Impulse Inhibition in Adolescents With Non-suicidal Self-injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Wang Meiling, student, Anhui Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AHMU-beta-band-tACS-NSSI
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Depression Disorders; Non-suicidal Self-injury
Keywords: Depression; non-suicidal self-injury; transcranial alternating current stimulation
MeSH Terms: conditions — Self-Injurious Behavior; Depression

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Active stimulation: deliver 20 minutes of beta-band tACS intervention.
  Interventions: Device: Beta-frequency transcranial alternating current stimulation
- Control group (Sham Comparator): Sham stimulation will be administered with identical treatment parameters, duration, and number of sessions as the active intervention. For the control group, the current will be ramped up to 2 mA and then ramped down to 0 mA within the first 30 seconds.
  Interventions: Device: sham beta-frequency transcranial alternating current stimulation

INTERVENTIONS:
Device: Beta-frequency transcranial alternating current stimulation — Active beta-frequency transcranial alternating current stimulation: 20 Hz tACS delivered through a 4×1-ring high-definition electrode montage centered on left DLPFC (F3), 2 mA peak-to-peak, 100 % intensity, gradually ramped up over 30 s, maintained for 20 min, then ramped down over 30 s; two sessions per day with at least 4 h between sessions, repeated for 7 consecutive days (14 total sessions).
  Arms: Experimental group
Device: sham beta-frequency transcranial alternating current stimulation — Sham transcranial alternating current stimulation: identical 4×1-ring high-definition electrode montage centered on left DLPFC (F3), 2 mA peak-to-peak current ramped up over 30 s and immediately ramped down to 0 mA, followed by 19.5 min of no stimulation to match the 20-min session duration of active tACS; delivered twice daily (≥4 h apart) for 7 consecutive days (14 total sessions).
  Arms: Control group

SUMMARY:
This clinical trial aims to determine whether beta-band transcranial alternating current stimulation (tACS) can improve impulse inhibition in adolescents with non-suicidal self-injury (NSSI) and to evaluate its safety. The primary questions it seeks to answer are:

* Can beta-band tACS significantly reduce the frequency of self-injury and scores on impulsivity scales in adolescents with NSSI?
* What discomfort or medical issues may participants experience during tACS intervention?

Researchers will compare beta-band tACS with sham stimulation (a procedure that mimics the real stimulation without delivering effective current) to verify its efficacy.

Participants will:

* Receive two sessions of either tACS or sham stimulation daily, spaced 4 hours apart, for 7 consecutive days (14 sessions in total).
* Undergo scale assessments, behavioral tasks, and eye-tracking tests before and after the intervention.
* Record any self-injury episodes and adverse reactions, with continuous monitoring and psychological support provided by a professional team.

ELIGIBILITY:
Inclusion Criteria:

* 1) Meet the proposed diagnostic criteria for non-suicidal self-injury (NSSI) in the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5), with ≥5 documented self-injury episodes and at least one incident within the past month as assessed by the Adolescent Non-Suicidal Self-Injury Assessment Questionnaire (ANSAQ); 2) Aged 12-18 years; 3) Right-handed; 4) Possess formal education experience sufficient to comprehend experimental protocols; 5) Normal or corrected-to-normal binocular visual acuity; 6) Voluntarily participate with legal guardians providing written informed consent.

Exclusion Criteria:

* 1) Montreal Cognitive Assessment (MoCA) score < 26; 2) History of suicide attempt(s); 3) Medical history of epilepsy, brain surgery, intracranial tumors, metal implants in the skull, or clinically significant head trauma; 4) History of substance use disorder, brain injury, severe somatic diseases, psychiatric disorders, or comorbid DSM-5 psychiatric conditions; 5) Prior receipt of transcranial direct current stimulation (tDCS), transcranial alternating current stimulation (tACS), or repetitive transcranial magnetic stimulation (rTMS) within the past 3 months

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Adolescent Non-suicidal Self-injury Assessment Questionnaire (ANSAQ) reduction in the frequency of self-injury | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The ANSAQ is a brief, self-report tool specifically designed for adolescents aged 12-18 to quantify non-suicidal self-injury (NSSI) over the past year. It is used both to screen for clinically relevant self-harm and to track changes in self-injury frequency after an intervention.
UPPS-P Impulsive Behavior Scale (UPPS-P) | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The UPPS-P is a 59-item self-report questionnaire that measures five distinct facets of impulsivity: Negative Urgency, (lack of) Premeditation, (lack of) Perseverance, Sensation Seeking, and Positive Urgency. Each item is rated on a 4-point Likert scale from 1 (agree strongly) to 4 (disagree strongly); items are reverse-scored so that higher scores indicate greater impulsivity.
Brief Barratt Impulsiveness Scale (BBIS) | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The BBIS is an 8-item, self-report subset of the well-known Barratt Impulsiveness Scale. Each item (e.g., "I act on the spur of the moment") is answered on a 4-point scale: 1 = rarely/never, 2 = occasionally, 3 = often, 4 = almost always/always. Total scores range 8-32; higher scores indicate greater impulsivity.
Eye movement index-fixation time | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  Recorded with an SMI-RED eye-tracker while participants freely view 60 pictures in the NSSI-cue reactivity paradigm. Each picture (tool cue, use cue, association cue, or neutral cue) is presented for 4 000 ms. The Region of Interest (ROI) is the entire picture area. "Fixation time" is the total duration (ms) that gaze remains within this ROI during picture presentation. Values are averaged across all cue types (or separately for NSSI-relevant vs. neutral cues) at baseline (Day 0) and post-intervention (Day 8). A ≥ 20 % reduction in total fixation time on NSSI-relevant cues relative to baseline is defined as a clinically relevant improvement in inhibitory control.
Eye movement index-fixation counts | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  During the NSSI cue-reactivity paradigm, an SMI-RED eye-tracker records gaze while 60 pictures (tool, use, association, or neutral cues) are each displayed for 4 000 ms. The entire picture is defined as the Region of Interest (ROI). "Fixation counts" is the total number of discrete fixations that fall within this ROI. The score is averaged across all pictures (or separately for NSSI-relevant vs. neutral cues) at baseline (Day 0) and after the 7-day intervention (Day 8). A ≥ 20 % reduction in fixation counts on NSSI-relevant cues from baseline indicates improved impulse inhibition.
Balloon Analog Risk Task-Total number of Balloon explosions | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  In the computer-based Balloon Analog Risk Task (BART), participants are shown 30 virtual balloons one at a time. They press "F" to inflate (pump) each balloon; every pump increases potential earnings by ¥0.5 but also raises the risk of explosion. Explosion points are random (1-128 pumps, mean 64). Participants can press "J" at any time to stop inflating and bank the current reward. "Total number of balloon explosions" is the count of balloons that burst across all 30 trials. Higher numbers reflect greater risk-taking and poorer impulse control. The score is obtained at baseline (Day 0) and after the 7-day intervention (Day 8); a ≥ 20 % reduction in explosions from baseline is considered a clinically relevant improvement in inhibitory control.

SECONDARY OUTCOMES:
Hamilton Depression Scale (HAMD-17) score | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The HAMD-17 is a clinician-rated scale of depressive symptoms. Seventeen items (mood, sleep, guilt, etc.) are scored 0-2 or 0-4; total ranges 0-52. Higher scores indicate more severe depression.
Hamilton Anxiety Scale (HAMA-14) score | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The HAMA-14 is a clinician-rated scale that assesses the severity of anxiety symptoms. It contains 14 items covering psychic and somatic anxiety; each item is scored 0 (not present) to 4 (very severe), giving a total range of 0-56, with higher scores indicating greater anxiety.
the score of Moca | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  A 30-point clinician-administered screen covering eight cognitive domains: visuospatial/executive, naming, memory, attention, language, abstraction, delayed recall, and orientation. Each correct response earns 1 point; scores 0-30 with ≥ 26 considered normal. Used in this study to exclude participants with cognitive impairment (< 26).
the score of TAS-20 | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  Self-report measure of alexithymia with 20 items rated 1-5, yielding three subscales: Difficulty Identifying Feelings, Difficulty Describing Feelings, and Externally Oriented Thinking. Total score 20-100; ≥ 61 indicates clinically significant alexithymia.
the score of ERQ | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  The ERQ is a 10-item self-report scale that measures habitual use of two emotion-regulation strategies: Cognitive Reappraisal (6 items) and Expressive Suppression (4 items). Each item is rated on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree). Sub-scale scores are generated by summing respective items: Reappraisal range 6-42, Suppression range 4-28. Higher scores indicate more frequent use of the strategy. The scale shows good internal consistency (α ≥ .79) and 3-month test-retest reliability (r ≈ .69) in adolescents .
the score of PANSI | Once at baseline (pre-treatment) and once at the end of treatment on Day 8.
  14-item self-report that gauges both protective (positive) and risk-related (negative) aspects of suicide ideation in adolescents. Items are rated 1-5; higher totals on the 6-item Positive Ideation sub-scale (range 6-30) indicate greater resilience, while higher totals on the 8-item Negative Ideation sub-scale (range 8-40) signal increased suicide risk.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, doctor, Study Director — School of Mental Health and Psychological Sciences, Anhui Medical University
Locations (1):
- School of Mental Health and Psychological Sciences, Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided